CLINICAL TRIAL: NCT05515588
Title: A Phase I, Open-label Trial to Investigate Metabolism, Pharmacokinetics (Following a Mass Balance Design) and Absolute Bioavailability of BI 690517 (C-14) After Oral and Intravenous Administration in Healthy Male Subjects
Brief Title: A Study in Healthy Men to Test How BI 690517 is Taken up and Handled by the Body
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1378-0013; 2022-001818-18 (EudraCT Number)
Record Dates: First submitted 2022-08-24; First posted 2022-08-25 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-09

CONDITIONS: Healthy
MeSH Terms: interventions — Carbon-14

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Part A: BI 690517 (C-14) (Experimental)
  Interventions: Drug: BI 690517 (C-14)
- Part B: BI 690517 fasted (test treatment, T) / BI 690517 (C-14) (reference treatment, R) (Experimental)
  Interventions: Drug: BI 690517 (C-14); Drug: BI 690517

INTERVENTIONS:
Drug: BI 690517 (C-14) — BI 690517 (C-14)
  Other Names: Vicadrostat
Drug: BI 690517 — BI 690517
  Other Names: Vicadrostat
  Arms: Part B: BI 690517 fasted (test treatment, T) / BI 690517 (C-14) (reference treatment, R)

SUMMARY:
The trial is intended to investigate the basic pharmacokinetics, excretion pathways and metabolism of BI 690517 and its metabolites.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects according to the assessment of the investigator, as based on a complete medical history including a physical examination, vital signs (Blood pressure (BP), Pulse rate (PR)), 12-lead Electrocardiogram (ECG), and clinical laboratory tests.
* Age of 18 to 55 years (inclusive).
* Body mass index (BMI) of 18.5 to 29.9 kg/m2 (inclusive).
* Signed and dated written informed consent in accordance with International Council for Harmonisation-Good Clinical Practice (ICH-GCP) and local legislation prior to admission to the trial.

Exclusion Criteria:

Subjects will not be allowed to participate, if any of the following general criteria apply:

* Any finding in the medical examination (including BP, PR or ECG) deviating from normal and assessed as clinically relevant by the investigator.
* Repeated measurement of systolic blood pressure outside the range of 90 to 140 millimetre(s) of mercury (mmHg), diastolic blood pressure outside the range of 45 to 90 mmHg, or pulse rate outside the range of 40 to 100 beats per minute (bpm).
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance.
* Any evidence of a concomitant disease assessed as clinically relevant by the investigator.
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders.
* Cholecystectomy or other surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy or simple hernia repair).
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders.
* History of relevant orthostatic hypotension (including but not limited to a reduction in systolic BP of ≥20 mm Hg or in diastolic BP of ≥10 mm Hg within 3 minutes of standing during screening measurement associated with clinical symptoms), fainting spells, or blackouts.

Further exclusion criteria apply.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2022-09-19 (Actual); Primary Completion 2022-11-17 (Actual); Study Completion 2022-11-17 (Actual)

PRIMARY OUTCOMES:
Part A: Fraction of [14C] radioactivity excreted into urine given as percentage of the administered dose in the time interval from 0 to last quantifiable time point (fe urine,0-tz ) | Up to 22 days.
Part A: Fraction of [14C] radioactivity excreted into feces given as percentage of the administered dose in the time interval from 0 to last quantifiable time point (fe feces, 0-tz) | Up to 22 days.
Part B: Area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity after intravenous administration (AUC0-∞) | Up to 3 days.
Part B: Area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity after oral administration (AUC0-∞) | Up to 3 days.

SECONDARY OUTCOMES:
Part A: Area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the last quantifiable time point (AUC0-tz) | Up to 8 days.
Part A: Maximum measured concentration of the analyte in plasma (Cmax) | Up to 8 days.
Part B: Maximum measured concentration of the analyte in plasma (Cmax) | Up to 3 days.
Part B: Area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the last quantifiable time point (AUC0-tz) | Up to 3 days.

CONTACTS AND LOCATIONS:
Locations (1):
- ICON, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to:
  https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com/